CLINICAL TRIAL: NCT01946789
Title: A Phase 1 Study of the Clinical and Immunologic Effects of ALT-803, a Novel Recombinant IL-15 Complex in Patients With Advanced Solid Tumors: Melanoma, Renal Cell, Non-Small Cell Lung and Squamous Cell Head and Neck Cancer
Brief Title: A Phase 1 Study of the Clinical and Immunologic Effects of ALT-803 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Altor BioScience (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CITN06-ALT-803, QUILT-3.003; U01CA154967 (NIH)
Record Dates: First submitted 2013-09-11; First posted 2013-09-20 (Estimated); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Advanced Solid Tumors
Keywords: cancer; IL-15; melanoma; metastatic; unresectable; solid tumors; renal cell; non-small cell lung; squamous cell head and neck
MeSH Terms: conditions — Neoplasms; Melanoma; Neoplasm Metastasis | interventions — ALT-803

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- N-803 IV 0.3/0.5 ug/kg (Experimental)
  Interventions: Biological: ALT-803
- N-803 IV 1.0 ug/kg (Experimental)
  Interventions: Biological: ALT-803
- N-803 IV 3.0 ug/kg (Experimental)
  Interventions: Biological: ALT-803
- N-803 IV 6.0 ug/kg (Experimental)
  Interventions: Biological: ALT-803
- N-803 Subcutaneous 6.0 ug/kg (Experimental)
  Interventions: Biological: ALT-803
- N-803 Subcutaneous 10.0 ug/kg (Experimental)
  Interventions: Biological: ALT-803
- N-803 Subcutaneous 15.0 ug/kg (Experimental)
  Interventions: Biological: ALT-803
- N-803 Subcutaneous 20.0 ug/kg (Experimental)
  Interventions: Biological: ALT-803
- N-803 Intratumoral 10.0 ug/kg followed by N-803 15.0 ug/kg subcutaneous (Experimental)
  Interventions: Biological: ALT-803

INTERVENTIONS:
Biological: ALT-803 — N-803 will be administered at the following doses intravenously: 0.3/0.5, 1.0, 3.0, 6.0 ug/kg N-803 will be administered at the following does subcutaneously: 6.0, 10.0, 15.0, 20.0 ug/kg N-803 will be administered intratumorally at a dose of 10.0 ug/kg, followed by N-803 administered subcutaneously at a dose of 15.0 ug/kg. Each treatment cycle consists of 4 weeks on therapy and 2 weeks off. Patients will receive weekly dose of ALT-803 for 4 weeks (Days 1, 8, 15, and 22) used for the identification of the OBD and MTD. After a 2-week rest period (Weeks 5 and 6) and recovery of any dose limiting toxicities to grade 0-1 of Cycle 1, a second 6-week cycle (4 weeks on treatment and 2 weeks off) can begin. After a rest period during Weeks 5 and 6 of Cycle 2, stable or benefitting patients assessed at week 8 +/- 1 may receive up to 2 additional 6-week cycles.

SUMMARY:
The proposed clinical trial is a phase I, open-label, multi-center, dose-escalation study of ALT-803 in patients with surgically incurable advanced solid tumors: melanoma, renal cell, non-small cell lung and squamous cell head and neck cancer

DETAILED DESCRIPTION:
This trial will investigate the safety and immunogenicity, immunomodulatory properties, and clinical benefits of treatment with weekly doses of ALT-803 in patients with advanced solid tumors.

ELIGIBILITY:
ENTRY CRITERIA:

DISEASE CHARACTERISTICS:

* Histological or cytological confirmed malignancy in the following disease groups: melanoma that is metastatic or unresectable, non-small cell lung carcinoma, renal cell carcinoma or squamous cell head and neck carcinoma, for which standard curative or palliative measures do not exist or are no longer effective.
* Primary site may be cutaneous or unknown, but mucosal and ocular primaries are excluded.
* Patients with non-small lung cancer must have had prior EGFR and ALK testing. Patients with sensitizing mutations in EGFR or ALK rearrangements should have been treated with prior targeted agents and have had progression or discontinued due to toxicity from these agents.
* No patients with known brain metastases.

PRIOR/CONCURRENT THERAPY:

* At least one prior therapy using an agent with the potential for prolonged remission.
* Patients with BRAF v600 mutation should be excluded or may be included after experiencing progression following treatment with BRAF inhibitor regimen or if they consent to forgo FDA-approved therapies that increase median survival.
* At least 4 weeks from last dose of prior chemotherapy or immunomodulator therapy with full recovery of acute toxicities. For patients coming off molecularly-targeted therapy, at least 2 weeks since last dose and recovery from laboratory and constitutional toxicities.
* At least 2 weeks from completion of prior radiation therapy with full recovery from toxicities.
* At least 4 weeks from last dose of prior investigational therapy with recovery to meet baseline eligibility criteria.
* Not receiving any current anticancer therapy
* No patients who have had chemotherapy, targeted therapy, or radiotherapy and have not recovered from acute toxicity to their pretreatment baseline or to a grade 1 level within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study. For resolution of autoimmune toxicity from prior immune therapy, patients must be off steroids for at least 30 days without relapse of autoimmune toxicity, or it must be at least 30 days from their last dose of infliximab or related immunosuppressive therapy without relapse of autoimmune toxicity.
* No patients who are receiving any other investigational agents.
* No patients who are receiving chronic systemic or regular inhaled corticosteroid use within 7 days prior to initiation of protocol therapy.
* No immunosuppressive therapy within 30 days prior to treatment start.

PATIENT CHARACTERISTICS

* Age >18 years
* Both men and women of all races and ethnic groups are eligible.

Performance Status

* ECOG performance status ≤1
* Life expectancy of greater than 6 months.

Bone Marrow Function

* leukocytes ≥3,000/mcL
* absolute lymphocyte count ≥500/mcL
* absolute neutrophil count ≥1,000/mcL (without hematopoietic growth factors)
* platelets ≥100,000/mcL (without transfusion)
* hemoglobin ≥ 10 gm/dL (may be transfused but must be stable without clinical evidence of ongoing blood loss or hemolysis)

Hepatic Function

* total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal

Kidney Function

* Creatinine within normal institutional limits OR
* Creatinine clearance ≥60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.

Pulmonary Function

• No history of severe COPD or emphysema or interstitial lung disease currently on home supplemental oxygen. Patients with NSCLC with stable COPD or emphysema not requiring supplemental oxygen are eligible.

Cardiac Function

* No symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia. Patients who have underlying risk factors for cardiac disease should be excluded or undergo clearance stress-based cardiac function testing. The pre-treatment QTc must be <500 msec.
* No class II or greater congestive heart failure as described in the New York Heart Association Functional Classification criteria or serious arrhythmias likely to increase the risk of cardiac complications of cytokine therapy.

Other

* Women of child-bearing potential and men must agree to use adequate contraception.
* Ability to understand and the willingness to sign a written informed consent document.
* No uncontrolled inter-current illness or psychiatric illness/social situations that would limit compliance with study requirements.
* No pregnant women.
* No HIV-positive patients.
* No positive hepatitis C serology or active hepatitis B infection.
* No active bacterial or fungal infection.
* No inability to home monitor blood pressure.
* Patients with thyroid disease should be excluded unless euthyroid on suppressive or replacement therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ernstoff, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (5):
- United States (5):
  - University of Minnesota, Minneapolis, Minnesota
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Washington, Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30045932/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | N-803 IV 0.3/0.5 ug/kg | N-803 IV 1.0 ug/kg | N-803 IV 3.0 ug/kg | N-803 IV 6.0 ug/kg | N-803 Subcutaneous 6.0 ug/kg | N-803 Subcutaneous 10.0 ug/kg | N-803 Subcutaneous 15.0 ug/kg | N-803 Subcutaneous 20.0 ug/kg | N-803 Intratumoral 10.0 ug/kg Followed by N-803 15.0 ug/kg Subcutaneous
Started | 2 | 3 | 3 | 3 | 3 | 3 | 4 | 3 | 2
Completed | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 0
Not Completed | 0 | 2 | 2 | 3 | 2 | 3 | 4 | 1 | 2
Not completed — Death | 0 | 2 | 1 | 1 | 1 | 1 | 3 | 1 | 2
Not completed — Progressive Disease | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N-803 IV 0.3/0.5 ug/kg | N-803 IV 1.0 ug/kg | N-803 IV 3.0 ug/kg | N-803 IV 6.0 ug/kg | N-803 Subcutaneous 6.0 ug/kg | N-803 Subcutaneous 10.0 ug/kg | N-803 Subcutaneous 15.0 ug/kg | N-803 Subcutaneous 20.0 ug/kg | N-803 Intratumoral 10.0 ug/kg Followed by N-803 15.0 ug/kg Subcutaneous | Total
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 3 | 4 | 3 | 2 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.0 (15.56) | 64.7 (6.81) | 58.7 (10.26) | 69.7 (8.02) | 59.3 (5.13) | 59.0 (3.46) | 63.3 (9.88) | 55.3 (10.97) | 64.0 (19.8) | 59.9 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2 | 1 | 1 | 1 | 3 | 1 | 0 | 11
  Male | 0 | 3 | 1 | 2 | 2 | 2 | 1 | 2 | 2 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 2 | 3 | 3 | 2 | 3 | 2 | 4 | 3 | 2 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 2 | 3 | 3 | 3 | 2 | 3 | 3 | 2 | 23
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Advanced Solid Tumors [Count of Participants; unit: Participants] | 2 | 3 | 3 | 3 | 3 | 3 | 4 | 3 | 2 | 26

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity
Description: The safety endpoint is the MTD of ALT-803, defined as the dose level below that at which ≥2 of 6 patients experience a DLT.
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | N-803 IV 0.3/0.5 ug/kg | N-803 IV 1.0 ug/kg | N-803 IV 3.0 ug/kg | N-803 IV 6.0 ug/kg | N-803 Subcutaneous 6.0 ug/kg | N-803 Subcutaneous 10.0 ug/kg | N-803 Subcutaneous 15.0 ug/kg | N-803 Subcutaneous 20.0 ug/kg | N-803 Intratumoral 10.0 ug/kg Followed by N-803 15.0 ug/kg Subcutaneous
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 3 | 4 | 3 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

2. Secondary Outcome: Number of Participants Who Developed Anti-drug Antibodies to ALT-803
Description: Immunogenicity of ALT-803 assessed by ELISA
Time Frame: 14 days post final dose, up to 135 days
Population: There were 2 participants in the N-803 IV 6.0 ug/kg, 1 participant in the N-803 Subcutaneous (SC) 6.0 ug/kg, and 1 participant in the N-803 Subcutaneous 20.0 ug/kg cohorts that had samples not collected. There were 2 subjects from the 6.0 ug/kg SC cohort whose samples were provided to the NantCell analytical laboratory and analyzed, but original assay reports could not be located and thus results cannot be reported.
Measure: Count of Participants; unit: Participants
Arm/Group | N-803 IV 0.3/0.5 ug/kg | N-803 IV 1.0 ug/kg | N-803 IV 3.0 ug/kg | N-803 IV 6.0 ug/kg | N-803 Subcutaneous 6.0 ug/kg | N-803 Subcutaneous 10.0 ug/kg | N-803 Subcutaneous 15.0 ug/kg | N-803 Subcutaneous 20.0 ug/kg | N-803 Intratumoral 10.0 ug/kg Followed by N-803 15.0 ug/kg Subcutaneous
Number analyzed (Participants) | 2 | 3 | 3 | 1 | 0 | 3 | 4 | 2 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: To Evaluate the Effect of Escalating Doses of ALT-803: Pharmacokinetics (Half Life and Tmax)
Description: Pharmacokinetics of ALT-803 assessed by ELISA
Time Frame: 24 hours post dose
Population: Results not available for each participant at each parameter because results were below the level of detection
Measure: Mean (Full Range); unit: hours
Groups:
- N-803 IV 0.3ug/kg; N-803 IV 1.0 ug/kg; N-803 IV 3.0 ug/kg; N-803 IV 6.0 ug/kg; N-803 Subcutaneous 6.0 ug/kg; N-803 Subcutaneous 10.0 ug/kg; N-803 Subcutaneous 15.0 ug/kg; N-803 Subcutaneous 20.0 ug/kg; N-803 Intratumoral 10.0 ug/kg Followed by N-803 15.0 ug/kg Subcutaneous; N-803 IV 0.5ug/kg: ALT-803: N-803 will be administered at the following doses intravenously: 0.3/0.5, 1.0, 3.0, 6.0 ug/kg N-803 will be administered at the following does subcutaneously: 6.0, 10.0, 15.0, 20.0 ug/kg N-803 will be administered intratumorally at a dose of 10.0 ug/kg, followed by N-803 administered subcutaneously at a dose of 15.0 ug/kg. Each treatment cycle consists of 4 weeks on therapy and 2 weeks off. Patients will receive weekly dose of ALT-803 for 4 weeks (Days 1, 8, 15, and 22) used for the identification of the OBD and MTD. After a 2-week rest period (Weeks 5 and 6) and recovery of any dose limiting toxicities to grade 0-1 of Cycle 1, a second 6-week cycle (4 weeks on treatment and 2 weeks off) can begin. After a rest period during Weeks 5 and 6 of Cycle 2, stable or benefitting patients assessed at week 8 +/- 1 may receive up to 2 additional 6-week cycles.
Arm/Group | N-803 IV 0.3ug/kg | N-803 IV 1.0 ug/kg | N-803 IV 3.0 ug/kg | N-803 IV 6.0 ug/kg | N-803 Subcutaneous 6.0 ug/kg | N-803 Subcutaneous 10.0 ug/kg | N-803 Subcutaneous 15.0 ug/kg | N-803 Subcutaneous 20.0 ug/kg | N-803 Intratumoral 10.0 ug/kg Followed by N-803 15.0 ug/kg Subcutaneous | N-803 IV 0.5ug/kg
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 1
hours
  Half life: number analyzed (Participants) | 1 | 2 | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 1
  Half life | 2.23 [2.23 to 2.23] | 4.58 [1.36 to 7.79] | 2.53 [2.53 to 2.53] | 1.41 [0.751 to 2.06] | NA [NA to NA] — below the level of detection | NA [NA to NA] — below the level of detection | NA [NA to NA] — below the level of detection | NA [NA to NA] — below the level of detection | 2.73 [2.3 to 3.15] | NA [NA to NA] — below the level of detection
  Tmax | 0.583 [0.583 to 0.583] | 0.542 [0.517 to 0.567] | 0.667 [0.533 to 0.8] | 0.650 [0.55 to 0.75] | 6.06 [4.0 to 8.12] | 24.0 [23.9 to 24.0] | 16.1 [8.0 to 24.3] | 16.1 [8.12 to 24.0] | 0.508 [0.5 to 0.517] | 0.500 [0.500 to 0.500]

4. Secondary Outcome: To Evaluate the Effect of Escalating Doses of ALT-803: Pharmacokinetics (Cmax)
Description: Pharmacokinetics of ALT-803 assessed by ELISA
Time Frame: 24 hours after first dose
Population: To Evaluate the Effect of Escalating Doses of ALT-803: Pharmacokinetics (Cmax). Results not available for each participant at each parameter because insufficient measurable concentration data.
Measure: Mean (Full Range); unit: ng/mL
Groups:
- N-803 IV 0.3 ug/kg; N-803 IV 1.0 ug/kg; N-803 IV 3.0 ug/kg; N-803 IV 6.0 ug/kg; N-803 Subcutaneous 6.0 ug/kg; N-803 Subcutaneous 10.0 ug/kg; N-803 Subcutaneous 15.0 ug/kg; N-803 Subcutaneous 20.0 ug/kg; N-803 Intratumoral 10.0 ug/kg Followed by N-803 15.0 ug/kg Subcutaneous; N-803 IV 0.5 ug/kg: ALT-803: N-803 will be administered at the following doses intravenously: 0.3/0.5, 1.0, 3.0, 6.0 ug/kg N-803 will be administered at the following does subcutaneously: 6.0, 10.0, 15.0, 20.0 ug/kg N-803 will be administered intratumorally at a dose of 10.0 ug/kg, followed by N-803 administered subcutaneously at a dose of 15.0 ug/kg. Each treatment cycle consists of 4 weeks on therapy and 2 weeks off. Patients will receive weekly dose of ALT-803 for 4 weeks (Days 1, 8, 15, and 22) used for the identification of the OBD and MTD. After a 2-week rest period (Weeks 5 and 6) and recovery of any dose limiting toxicities to grade 0-1 of Cycle 1, a second 6-week cycle (4 weeks on treatment and 2 weeks off) can begin. After a rest period during Weeks 5 and 6 of Cycle 2, stable or benefitting patients assessed at week 8 +/- 1 may receive up to 2 additional 6-week cycles.
Arm/Group | N-803 IV 0.3 ug/kg | N-803 IV 1.0 ug/kg | N-803 IV 3.0 ug/kg | N-803 IV 6.0 ug/kg | N-803 Subcutaneous 6.0 ug/kg | N-803 Subcutaneous 10.0 ug/kg | N-803 Subcutaneous 15.0 ug/kg | N-803 Subcutaneous 20.0 ug/kg | N-803 Intratumoral 10.0 ug/kg Followed by N-803 15.0 ug/kg Subcutaneous | N-803 IV 0.5 ug/kg
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 1
ng/mL | 91.2 [91.2 to 91.2] | 11.5 [10.2 to 12.8] | 49.8 [39.9 to 59.6] | 86.0 [79.0 to 93.0] | 0.276 [0.152 to 0.401] | 0.352 [0.290 to 0.413] | 0.685 [0.443 to 0.928] | 0.280 [0.252 to 0.307] | 72.6 [26.5 to 119] | 2.26 [2.26 to 2.26]

5. Secondary Outcome: To Evaluate the Effect of Escalating Doses of ALT-803: Pharmacokinetics (AUC 0-t, AUC0-24, AUC0-infinity)
Description: Pharmacokinetics of ALT-803 assessed by ELISA
Time Frame: 24 hours after first dose
Population: Results not available for each participant at each parameter because results were below the level of detection.
Measure: Mean (Full Range); unit: hr*ng/mL
Arm/Group | N-803 IV 0.3ug/kg | N-803 IV 1.0 ug/kg | N-803 IV 3.0 ug/kg | N-803 IV 6.0 ug/kg | N-803 Subcutaneous 6.0 ug/kg | N-803 Subcutaneous 10.0 ug/kg | N-803 Subcutaneous 15.0 ug/kg | N-803 Subcutaneous 20.0 ug/kg | N-803 Intratumoral 10.0 ug/kg Followed by N-803 15.0 ug/kg Subcutaneous | N-803 IV 0.5ug/kg
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 1
hr*ng/mL
  AUC 0-t | 236 [236 to 236] | 14.7 [10.5 to 18.8] | 105 [65.2 to 145] | 289 [186 to 392] | 4.66 [2.74 to 6.59] | 5.19 [4.86 to 5.51] | 10.9 [8.67 to 13.2] | 4.57 [3.73 to 5.41] | 323 [82.1 to 565] | NA [NA to NA] — below the level of detection
  AUC0-24: number analyzed (Participants) | 1 | 2 | 1 | 2 | 1 | 1 | 2 | 2 | 2 | 1
  AUC0-24 | 236 [236 to 236] | 14.7 [10.6 to 18.8] | 145 [145 to 145] | 290 [187 to 393] | 2.73 [2.73 to 2.73] | 4.86 [4.86 to 4.86] | 10.9 [8.56 to 13.2] | 4.56 [3.73 to 5.4] | 323 [82.1 to 564] | NA [NA to NA] — below the level of detection
  AUC0-infinity: number analyzed (Participants) | 1 | 2 | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 1
  AUC0-infinity | 236 [236 to 236] | 15.0 [10.5 to 19.4] | 145 [145 to 145] | 290 [187 to 393] | NA [NA to NA] — below the level of detection | NA [NA to NA] — below the level of detection | NA [NA to NA] — below the level of detection | NA [NA to NA] — below the level of detection | 324 [82.4 to 565] | NA [NA to NA] — below the level of detection

6. Secondary Outcome: To Evaluate the Effect of Escalating Doses of ALT-803: Interferon Gamma (IFN-γ)
Description: The level of immune response to autochthonous viral and tumor antigens by interferon gamma (IFN-γ) ELISPOT
Time Frame: Cycle 1 Week 1, pre-dose; Cycle 1 Week 1, 30 minutes post dose; Cycle 1 Week 1, 2 hours post dose; Cycle 1 Week 1, 4 hours post dose; Cycle 1 Week 1, 8 hours post dose; Cycle 1 Week 1, 24 hours post dose
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | N-803 IV 0.3/0.5 ug/kg | N-803 IV 1.0 ug/kg | N-803 IV 3.0 ug/kg | N-803 IV 6.0 ug/kg | N-803 Subcutaneous 6.0 ug/kg | N-803 Subcutaneous 10.0 ug/kg | N-803 Subcutaneous 15.0 ug/kg | N-803 Subcutaneous 20.0 ug/kg | N-803 Intratumoral 10.0 ug/kg Followed by N-803 15.0 ug/kg Subcutaneous
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 3 | 4 | 3 | 2
pg/mL
  C1, W1 pre dose | 2.7 (0.5037) | 1.528 (2.1609) | 2.015 (2.8496) | 0 (0) | 0.326 (0.3833) | 2.741 (2.3792) | 2.659 (4.6059) | 4.445 (7.6987) | 5.955 (0.5356)
  C1, W1 30min post dose | 0 (0) | 3.433 (4.8551) | 1.420 (2.0082) | 0 (0) | 0.163 (0.2829) | 0.692 (1.1994) | 2.659 (4.6059) | 1.394 (2.4152) | 2.397 (3.3896)
  C1, W1 2 hr post dose | 21.827 (25.6506) | 22.585 (2.9941) | 30.605 (36.7908) | 10.198 (13.8527) | 0 (0) | 1.525 (1.3373) | 0 (0) | 1.463 (2.5342) | 43.863 (42.2211)
  C1, W1 4 hr post dose | 64.947 (85.0197) | 47.160 (37.1485) | 57.660 (56.4978) | 23.295 (28.1061) | 1.146 (1.7892) | 1.771 (2.2307) | 0.607 (1.0506) | 1.325 (2.2943) | 78.729 (63.0940)
  C1, W1 8 hr post dose | 10.022 (14.1731) | 11.158 (4.7186) | 15.3 (9.8995) | 7.597 (9.5858) | 0 (0) | 2.123 (1.1098) | 2.479 (4.2939) | 1.598 (2.7676) | 22.293 (11.2426)
  C1, W1 24 hr post dose | 0 (0) | 0.728 (1.0292) | 0.73 (1.0324) | 0 (0) | 0.84 (0.7962) | 3.825 (0.5214) | 4.389 (7.6013) | 1.664 (2.8823) | 4.078 (5.7676)

7. Secondary Outcome: Objective Response Rate
Description: Number of patients with CR, PR, SD, and PD
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | N-803 IV 0.3/0.5 ug/kg | N-803 IV 1.0 ug/kg | N-803 IV 3.0 ug/kg | N-803 IV 6.0 ug/kg | N-803 Subcutaneous 6.0 ug/kg | N-803 Subcutaneous 10.0 ug/kg | N-803 Subcutaneous 15.0 ug/kg | N-803 Subcutaneous 20.0 ug/kg | N-803 Intratumoral 10.0 ug/kg Followed by N-803 15.0 ug/kg Subcutaneous
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 2 | 3 | 4 | 2 | 2
Participants
  Stable disease | 2 | 1 | 2 | 0 | 2 | 0 | 3 | 0 | 1
  Progressive disease | 0 | 2 | 1 | 3 | 0 | 3 | 1 | 2 | 1

ADVERSE EVENTS:
Time Frame: Up to 385 days.
Arm/Group | N-803 IV 0.3/0.5 ug/kg | N-803 IV 1.0 ug/kg | N-803 IV 3.0 ug/kg | N-803 IV 6.0 ug/kg | N-803 Subcutaneous 6.0 ug/kg | N-803 Subcutaneous 10.0 ug/kg | N-803 Subcutaneous 15.0 ug/kg | N-803 Subcutaneous 20.0 ug/kg | N-803 Intratumoral 10.0 ug/kg Followed by N-803 15.0 ug/kg Subcutaneous
All-Cause Mortality (participants affected / at risk) | 0/2 | 2/3 | 1/3 | 1/3 | 1/3 | 1/3 | 3/4 | 1/3 | 2/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/3 | 1/3 | 1/3 | 0/3 | 1/3 | 2/4 | 2/3 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 4/4 | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | N-803 IV 0.3/0.5 ug/kg (N=2) | N-803 IV 1.0 ug/kg (N=3) | N-803 IV 3.0 ug/kg (N=3) | N-803 IV 6.0 ug/kg (N=3) | N-803 Subcutaneous 6.0 ug/kg (N=3) | N-803 Subcutaneous 10.0 ug/kg (N=3) | N-803 Subcutaneous 15.0 ug/kg (N=4) | N-803 Subcutaneous 20.0 ug/kg (N=3) | N-803 Intratumoral 10.0 ug/kg Followed by N-803 15.0 ug/kg Subcutaneous (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | N-803 IV 0.3/0.5 ug/kg (N=2) | N-803 IV 1.0 ug/kg (N=3) | N-803 IV 3.0 ug/kg (N=3) | N-803 IV 6.0 ug/kg (N=3) | N-803 Subcutaneous 6.0 ug/kg (N=3) | N-803 Subcutaneous 10.0 ug/kg (N=3) | N-803 Subcutaneous 15.0 ug/kg (N=4) | N-803 Subcutaneous 20.0 ug/kg (N=3) | N-803 Intratumoral 10.0 ug/kg Followed by N-803 15.0 ug/kg Subcutaneous (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry Eye (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 0 | 1 | 1 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 2
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 1 | 2 | 1 | 0 | 3 | 3 | 1 | 2
Hypothermia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 4 | 3 | 2
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 1 | 1 | 2 | 1 | 1 | 2
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stoma site erythema (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Blood creatinine decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Blood iron decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Central nervous system lesion (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin discomfort (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-08-09): https://cdn.clinicaltrials.gov/large-docs/89/NCT01946789/Prot_000.pdf
  • Statistical Analysis Plan (2016-08-09): https://cdn.clinicaltrials.gov/large-docs/89/NCT01946789/SAP_001.pdf